CLINICAL TRIAL: NCT07273097
Title: Effects of Ankle Evertor Fatigue on Gait Perturbation Responses in Individuals With and Without Chronic Ankle Instability
Brief Title: Effects of Ankle Evertor Fatigue on Perturbed Gait
Status: Recruiting | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Alan Kacin, Head of Laboratory, University of Ljubljana
Other Study IDs: 0120-197/2023/3/gait
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: perturbed walking; fatigue; treadmill
MeSH Terms: conditions — Fatigue | interventions — Muscle Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Healthy participants without a history of ankle sprain or self-reported ankle instability. Participants in this group will complete the same experimental protocol as Chronic ankle instability group, which includes treadmill walking at two speeds (0.4 m/s and 1.0 m/s) with and without mechanical perturbations, performed before and after an ankle evertor fatigue protocol. For this group, the fatigued limb will be assigned based on the laterality of ankle sprains observed in the CAI group.
  Interventions: Other: Muscle fatigue
- Chronic ankle instability group: Participants with chronic ankle instability, defined by a history of recurrent ankle sprains and self-reported instability. Participants in this group will complete the same experimental protocol as Healthy group, which includes treadmill walking at two speeds (0.4 m/s and 1.0 m/s) with and without mechanical perturbations, performed before and after an ankle evertor fatigue protocol. For this group, the fatigued limb will be the symptomatic side.
  Interventions: Other: Muscle fatigue

INTERVENTIONS:
Other: Muscle fatigue — The fatigue protocol will consist of repeated concentric-eccentric ankle eversion contractions against elastic resistance at a pace of one repetition per second, guided by a metronome, and performed in a seated position. Fatigue will be defined as a clear inability to perform the full range of eversion, i.e. the range of motion falling below 50% of the initial value despite evident effort by the participant.

SUMMARY:
This study will investigate the effects of ankle evertor muscle fatigue on gait stability during treadmill walking with mechanical perturbations. Participants will walk at two speeds (0.4 m/s and 1.0 m/s) while random medial and lateral perturbations (<10% body weight) are applied to the pelvis. Surface EMG from ankle muscles and center of pressure (COP)-based gait parameters (e.g., step length, step width, single support duration, COP trajectory) will be analyzed before and immediately after an isotonic fatigue protocol of the ankle evertors.

DETAILED DESCRIPTION:
The purpose of this study is to examine how ankle evertor muscle fatigue affects gait stability and neuromuscular responses during treadmill walking with mechanical perturbations. Perturbations will be applied randomly in the medial or lateral direction, but always shortly after initial foot contact, to specifically challenge ankle stabilization in stance.

The study will include individuals with chronic ankle instability (CAI) and matched healthy controls. In the CAI group, the symptomatic side will be targeted with the fatigue protocol, whereas in healthy controls the tested side will be assigned to match the distribution of sprain laterality in the CAI group.

Walking and perturbation protocol:

Participants will first complete familiarization at 1.0 m/s, including both normal and perturbed walking. After familiarization, the measurements will consist of 2 minutes of unperturbed walking followed by 3 minutes of perturbed walking. The same procedure will then be repeated at 0.4 m/s, with familiarization (normal and perturbed walking) preceding the measurement block.

The fatigue protocol will be applied immediately after these baseline blocks. Following fatigue, participants will immediately perform perturbed walking at 1.0 m/s. The fatigue protocol will then be repeated, followed by perturbed walking at 0.4 m/s.

Fatigue protocol:

Ankle evertor muscles will be fatigued using elastic resistance bands through repeated concentric and eccentric eversion contractions. The task will be paced using a metronome at a rate of one repetition per second, and will continue until the active eversion range of motion decreases by 50% compared to baseline.

ELIGIBILITY:
Inclusion criteria for the healthy control group (no CAI):

* Age between 18 and 45 years,
* No history of injuries or surgical procedures to the lower limbs,
* No peripheral or central neurological impairments.

Inclusion criteria for the chronic ankle instability (CAI) group:

* Age between 18 and 45 years,
* No history of major surgical procedures on the lower limbs
* No peripheral or central neurological impairments,
* Diagnosed chronic ankle instability:

  * First ankle sprain occurred at least one year prior to testing,
  * At least three months since the most recent ankle sprain,
  * Subjective feeling of ankle instability - CAIT (Cumberland Ankle Instability Tool) score < 24.

Exclusion criteria for the CAI group:

* Other pathologies of the ankle joint.
* Acute pain

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited by convenience sampling from the general population and clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Surface EMG root mean square (RMS) amplitude of ankle muscles | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Surface EMG RMS amplitude from peroneus longus (PL), tibialis anterior (TA), soleus (SOL), gastrocnemius medialis (GM), and gluteus medius (GMed), recorded bilaterally during treadmill walking. EMG will be time-normalized to the gait cycle (0-100%). The primary epoch is the perturbation step (shortly after initial contact through stance). For each muscle and speed, EMG during perturbed walking will be normalized to matched unperturbed walking.
Center of Pressure mediolateral displacement (COPx) | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Mediolateral displacement of the center of pressure (COPx) during walking, time-normalized to the gait cycle (0-100%). In addition, COPx will be expressed relative to the sacral marker (COPx-SACRx). Values will be presented in absolute units (cm) and compared between matched perturbed steps at the same walking speed (before and after fatigue).

SECONDARY OUTCOMES:
Step Length and width | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Step length (heel-to-heel) and step width of the perturbation step, derived from 3D motion capture with reflective markers placed on anatomical landmarks. Both parameters will be compared against matched unperturbed steps.
Ground reaction forces (GRF) | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Vertical GRF (Fz; peak, mean, loading rate), with optional analysis of anteroposterior (Fy) and mediolateral (Fx) components, time-normalized to the gait cycle (0-100%). Values reported in absolute units (N for forces; N/s for loading rate).
Ratings of perceived exertion | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Description: Ratings of perceived exertion (RPE) will be assessed at the end of each fatigue protocol using the Borg 10 category-ratio scale, with 0 is no effort and 10 is an extreme physical effort.

CONTACTS AND LOCATIONS:
Locations (1):
- University Rehabilitation Institute Republic of Slovenia - URI Soča, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD in anonymized form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No limit.
Access Criteria: All IPD will be shared upon reasoned request for the purpose of further scientific analysis (i.e. systematic reviews, meta-analyzes, etc.). A proposal describing the planned analyzes must be submitted in writing to the principal investigator, Dr. Alan Kacin, by email to alan.kacin@zf.uni-lj.si.